CLINICAL TRIAL: NCT00342225
Title: Mother-Child Relationships During Pregnancy Among the Bofi Foragers in the Northern Congo
Brief Title: Mother-Child Relationships During Pregnancy Among Bofi Foragers
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903073; 03-CH-N073
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2006-12-21

CONDITIONS: Behavior
Keywords: Observation; Mothers; Description
MeSH Terms: conditions — Behavior

SUMMARY:
This study will examine changes in mother-child relationships when mothers are pregnant, because this period may involve conflicts between mothers and children. A widely held evolutionary theory postulates that because parents and offspring share only about 50 percent of their genes, conflicts occur and would most likely occur at times when parental investment decreases. Offspring benefit from obtaining maximal parental investment and may demand more investment than parents are willing to give at times, perhaps because the parent would better benefit from directing their energy to other pursuits, such as to other offspring or to work. This study will explore the following:

* How pregnant mothers treat their children, in terms of caregiving techniques;
* Whether mothers exhibit different caregiving patterns at different stages of pregnancy;
* Whether mother-child conflicts arise during pregnancy, and, if so, when during pregnancy they are most likely to occur; and;
* Whether offspring overtly resist changes in maternal behavior during pregnancy, and, if so, what behaviors children use to resist these changes.

All pregnant Bofi forager women living in settlements near the villages of Ngotto, Poutem, Bambondji, and Grima (in the Central African Republic) who have one or more living offspring and have no serious health problems related to pregnancy may be eligible for this study. Bofi foragers are among the few remaining hunters and gatherers and, as such, offer an opportunity to examine child developmental theories that have been well studied among industrialized Euro-American cultures, but neglected cross-culturally. Furthermore, studies among contemporary hunter-gatherers provide insight into the evolutionary past of humans, as humans have lived as hunter-gatherers for about 99 percent of prehistory.

Participating pregnant Bofi forager women will be interviewed for demographic information, family genealogy, fertility history, and parenting beliefs. The women and their children will be observed for 4 hours on two different days as they carry out their normal daily activities. Attention will be paid to the mother's investment in terms of direct care of the children, including behaviors such as holding, cleaning, comforting, grooming, and feeding children.

DETAILED DESCRIPTION:
This study seeks to examine parent-offspring reproductive conflicts between Bofi forager mothers and children in the Republic of Congo. One of the most prominent theories in evolutionary studies of human behavior is Trivers' (1974) parent-offspring conflict theory, which predicts that offspring contrive to maximize investment from their parents, whereas parents try to balance the interests of their offspring with the interests of their future reproduction. Fouts (2002) and Fouts, Hewlett & Lamb's (2001) research with the Bofi foragers indicated that weaning was not a time that elicited overt conflict between mothers and their offspring. Instead, transitions in investment appeared to have occurred prior to weaning, perhaps when the mothers became pregnant.

This study proposes to document mother-child interactions when forager mothers are at different stages of pregnancy through naturalistic observations of public behavior, as well as measures including: the approximate week of pregnancy, maternal beliefs about child-care, and demographic features of families. The data will be analyzed statistically and used to evaluate Trivers' parent-offspring theory, as well as to evaluate the validity of claims by Western scholars about universal features of parent-child relationships. The foragers provide an excellent opportunity to examine child developmental theories that have been well studied among industrialized Euro-American cultures, but neglected cross-culturally. Furthermore, studies among contemporary hunter-gatherer groups, such as the foragers in Congo, provide insight into the evolutionary past of humans, as humans have lived as hunter-gatherers for approximately 99% of prehistory, and the few remaining groups are disappearing rapidly (Phillipson 1993).

ELIGIBILITY:
* INCLUSION AND EXCLUSION CRITERIA:

All pregnant forager women living in settlements associated with the villages of Ouesso, Kobu, and Bomassa, who have one or more living offspring, and do no exhibit any serious health problems related to pregnancy will be asked to participate. Women will not be excluded based upon economic or social status, marital status, or spiritual beliefs.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2002-12-19; Study Completion 2006-12-21

CONTACTS AND LOCATIONS:
Locations (2):
- Central African Republic (2):
  - Central African Republic, Ngotto
  - Republic of Condo, Sangha

REFERENCES:
- [Background] Hewlett BS, Lamb ME, Shannon D, Leyendecker B, Scholmerich A. Culture and early infancy among central African foragers and farmers. Dev Psychol. 1998 Jul;34(4):653-61. doi: 10.1037//0012-1649.34.4.653. PMID 9681257